CLINICAL TRIAL: NCT03539874
Title: Impact of Sperm Oxidative Stress on Embryonic Parameters and Pregnancy Success During Intrauterine Insemination and in Vitro Fertilization
Brief Title: Sperm Oxidative Stress and Pregnancy Success During IUI and IVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fertilys (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-01
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sperm sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Confirmed paternity: Sperm sample from men with confirmed paternity
- Intrauterine insemination: Sperm sample from men in intrauterine insemination process
- In vitro fertilization: Sperm sample from men in in vitro fertilization process

SUMMARY:
Oxidative stress (OS) is characterized by an imbalance between the production of reactive oxygen species (ROS) and the ability of the body to eliminate them. Such an imbalance can lead to lipid peroxidation, DNA damage and cell apoptosis. Studies have suggested that infertile men are more likely to have high concentrations of ROS in their seminal plasma. The investigators hypothesize that a high level of oxidative stress (OS) in patients with abnormal sperm parameters could influence fertilization and / or pregnancy success. Our first goal is to compare OS levels to semen parameters, as defined by the World Health Organization in 2010, as well as DNA fragmentation and chromatin decondensation in sperm. Our second objective is to compare OS levels in sperm to fertilization and blastulation rates at first, and then measure the impact of OS levels on pregnancy success, both in intrauterine insemination (IUI) and in vitro fertilization (IVF). Sperm samples from men in 3 groups will be analyzed: a group of fertile men with confirmed paternity (n = 50), a group of men in IVF (n = 100) and a group of men in their first three cycles of IUI (n = 100). The static oxidation reduction index (sORP) will be measured by the MiOXSYS © system, a rapid sperm analysis system using electrochemical technology. A small portion of the fresh sperm sample will be deposited on a MiOXSYS sensor and the ORP will be measured. Sperm ROS will also be measured using the CellROX Deep Red probe. The sperm parameters will be measured by the techniques used routinely in the Fertilys Reproductive Health Center andrology lab. Regarding couples in IVF, fertilization and blastulation rates, embryo quality and pregnancy success will be noted. Pregnancy success will be noted for IUI couples. If the usefulness of sORP levels in predicting pregnancy and its outcome is demonstrated, it could be a new marker in the diagnosis of male infertility and act as a guide for clinicians to apply appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

* All men with confirmed paternity aged 18 to 40 years, agreeing to participate in the study and having signed the consent form.
* All patients aged 18 to 40 using IVF or their first cycle of IUI at the Fertilys Reproductive Health Center, agreeing to participate in the study and having signed the consent form.

Exclusion Criteria:

* Patients under 18 and over 40 years old.
* Men who can not produce a sperm sample by anterograde ejaculation.
* Men going to the Fertilys Reproductive Health Center for a post-vasectomy spermogram.
* Couples who have already completed IUI cycles.
* Couples using gamete donation (eggs or sperm).
* Men with a mobile sperm concentration of less than 5 millions/mL after preparation of the sperm sample during the IUI process.

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: All patients aged 18-40 in their first IUI cycle or IVF at the Fertilys Reproductive Health Center.
  All men whose paternity is confirmed who come to the Fertilys Reproductive Health Center for a spermogram.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Static oxidation reduction potential | 1 year
  Electrical measure given by the MiOXSYS System
Reactive Oxygen Species levels | 1 year
  Reactive Oxygen Species levels in sperm using the CellRox Deep Red probe

SECONDARY OUTCOMES:
Fertilization and blastulation rates | 1 year
  Fertilization and blastulation rates compare to the sperm oxidative stress levels
Pregnancy success | 1 year
  Pregnancy outcome in IUI and IVF according to sperm oxidative stress levels

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claire Bélanger, PhD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- Fertilys, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided